CLINICAL TRIAL: NCT01853332
Title: Physical Health in Midlife: Influences of Adversity and Relationships Over Time
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Judge Baker Children's Center (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Christos Mantzoros, Professor of Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2008P000424; R01AG032030 (NIH)
Record Dates: First submitted 2013-04-30; First posted 2013-05-15 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Disease; Type 2 Diabetes
Keywords: Cardiovascular Disease; Diabetes; Adjustment; Adversity; Psychology; Midlife; Functioning; Socioeconomic; Psychosocial outcomes
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and plasma are stored to be analyzed for biomarkers related to metabolic syndrome.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cross-Sectional: New participant: The purpose of the study is to learn about physical health in midlife and how it has been influenced by experiences and relationships. The study specifically targets health differences and the development of heart disease and diabetes.
- Longitudinal: Former participants (or the partner of a former participant) of the Adolescent and Family Development Project, Young Adult Development Project, Across Generations Project, and/or Paths Over Time Project may already know that this research shows how people grow, individually and as part of a familial and social network, throughout the course of life. This study focuses on learning about former participants' physical health in midlife and how it has been influenced by their experiences and relationships.

SUMMARY:
The purpose of this study is to determine the effects of individual characteristics, life stresses, and relationships over time on psychosocial outcomes (e.g. marriage, parenting, work) and physical health

DETAILED DESCRIPTION:
Research Procedures: If a patient choose to take part in this research study, they will undergo these research procedures:

The patient will participate in a total of two meetings and four phone calls over the course of the study (two and a half years). The meetings will be held at the beginning and end of the two and a half year period. The first part of each meeting will take place at Beth Israel Deaconess Medical Center (BIDMC) where they will sign this consent form and then be interviewed for medical history, given a physical examination, and have blood tests described below. The patient will then be transported to Judge Baker Children's Center (JBCC), where they will have lunch, complete questionnaires, and participate in taped interviews (approximately 4 hours). The phone calls will be approximately every six months and the patient will be contacted by the people at JBCC. More detailed information on the study procedures is outlined below and on the JBCC consent form for the study.

Interviews, Questionnaires, and Phone calls: These aspects of the study are covered in the Judge Baker Children's Center consent form. Briefly, the patient will be asked to discuss relationships with their partner, family, and friends, their career, their current goals in life, their health status, etc. These sessions will be recorded so that the patient's answers can be coded and analyzed at a later time. All information will be kept strictly confidential.

Medical Examination: The patient will arrive fasting to the medical examination. During the medical exam, a physician will ask the patient questions about their physical health and family history. The doctor will then conduct a physical examination which includes:

1. Glucose finger stick for diabetes screening
2. Vital signs (such as blood pressure) and anthropometrics (such as waist circumference).
3. Measuring the amount of fat in the patient's body using bioelectrical impedance analysis. This test will measure the resistance to the naturally occurring flow of electrical currents within the nerves and muscles using a few electrical sensors (similar to the EKG) attached to the patient's wrist and ankle for less than a minute. This procedure is not painful and uses the same principle as weighing oneself on a scale that provides body mass index.
4. Measuring the patient body's ability to use sugar through an oral glucose tolerance test (OGTT). A nurse will place an intravenous (IV) catheter (a small tube) in the patient's arm. It will be taped to stay in place for approximately four hours. The patient will drink a mixed nutrient drink called Boost. The patient's blood will be drawn through the catheter 15 min after the Boost is given and then at 30-minute intervals for 3 hours to measure how they metabolize the nutrient drink.
5. EKG

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between 35 and 55 years of age.

Exclusion Criteria: (based on interference with key assessments)

* Abnormal hepatic function (liver function tests >2X upper normal);
* abnormal renal function (creatinine >1.3 mg/dl);
* conditions/illnesses such as active infection, significant malabsorption/malnutrition, cancer;
* active hormonal disease such as overt hypo/hyperthyroidism, hypogonadism, hyper-cortisolism, or treatment with steroids or growth hormone.
* Known Diabetes Mellitus (DM) and Cardiovascular Disease (CVD) will be screened for by a detailed history and systems review.
* Baseline laboratory analysis with chemistries, CBC, hormone levels, and EKG will be completed.

Two exceptions will be made to the usual exclusion criteria:

1. Original subjects with DM or CVD will not be excluded, since that would result in bias in that sample and loss of opportunity to examine predictors associated with these outcomes.
2. Community adults diagnosed with these disorders at the screening visit will be retained and referred for medical treatment as needed. In both groups, those with DM and/or CVD will be followed for psychosocial and relevant biomedical variables, excluding assessments interfered with by CVD and DM relevant medications. Those with DM and CVD will at times be separately analyzed, together with participants who develop these disorders in the years of this new study phase.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Approximately 165 former participants and 250 new participants will take part in this study at Beth Israel Deaconess Medical Center (and Judge Baker Children's Center). The new sample will include 250 African American and Black Caribbean midlife men and women with the goal of recruiting 80% as couples. A total of 415 people will take part in this study at all study sites. Spouses and long-term significant others (with bonuses to couples for joining) will be encourage to also participate in the study. Targeting couples in this way will be parallel for the community and longitudinal samples
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2009-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos Mantzoros, MD, DSc, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Judge Baker Children's Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ko BJ, Park KH, Shin S, Zaichenko L, Davis CR, Crowell JA, Joung H, Mantzoros CS. Diet quality and diet patterns in relation to circulating cardiometabolic biomarkers. Clin Nutr. 2016 Apr;35(2):484-490. doi: 10.1016/j.clnu.2015.03.022. Epub 2015 Apr 7. PMID 25912185

RESULTS

PARTICIPANT FLOW:
Groups:
- Cross-Sectional: New participants: The purpose of the study is to learn about physical health in midlife and how it has been influenced by experiences and relationships. The study specifically targets health differences and the development of heart disease and diabetes.
  AND
  Former participants (or the partner of a former participant) of the Adolescent and Family Development Project, Young Adult Development Project, Across Generations Project, and/or Paths Over Time Project may already know that this research shows how people grow, individually and as part of a familial and social network, throughout the course of life. This study focuses on learning about former participants' physical health in midlife and how it has been influenced by their experiences and relationships.
Period: Overall Study
Arm/Group | Cross-Sectional
Started | 210
Completed | 151
Not Completed | 59

BASELINE CHARACTERISTICS:
Groups:
- Cross-Sectional: New and Former Participants
Arm/Group | Cross-Sectional
Number analyzed (Participants) | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 75

OUTCOME MEASURES:

1. Primary Outcome: Hormonal Levels
Description: To assess clinically significant physical health outcomes including 1) establishing risk factors for CVD and type 2 diabetes mellitus (DM) 2) establishing novel risk factors for CVD and DM (e.g., inflammatory markers, hormonal mediators ), and 3) determining the prevalence of established CVD and DM.
  1. Both insulin and glucose will be measured.
  2. Adipokines.
  3. Myokines.
  4. Triglycerides and HDL cholesterol will be considered in light of their relevance to CVD.
  5. Proinflammatory markers.
Time Frame: 2.5 years
Measure: Mean (Inter-Quartile Range); unit: ng/ml
Groups:
- Cross-Sectional: New participants and former participants
Arm/Group | Cross-Sectional
Number analyzed (Participants) | 151
ng/ml
  glucose | 910000 [840000 to 960000]
  insulin | 5.8 [3.2 to 10.3]
  adipokines (leptin) | 22.8 [6.9 to 37.0]
  myokines (irisin) | 171.8 [142.5 to 214.2]
  triglycerides | 820000 [600000 to 1170000]
  HDL-cholesterol | 530000 [450000 to 650000]
  proinflammatory markers (CRP) | 16000 [6000 to 37000]

2. Primary Outcome: Psychosocial Adversity
Description: Cumulative adversity occurring before age 18 was assessed using a) the Evaluation of Lifetime Stressors, b) SCID, and c) the Adult Attachment Interview. A cumulative adversity sum score was obtained (range 0-13, higher more).An overall adversity score was created by multiplying the number of childhood adversities×the overall severity of childhood adversity × the overall chronicity of childhood adversity. Scores for overall adversity ranged from 0 (no) to 156 more adversity).The Social Adjustment Scale is a semi-structured interview assessing functioning in the preceding 2 months and ranges from 1 (excellent) to 7 (very poor adjustment). An index score of psychosocial risk factors was created. Education less than a Bachelor's degree, unemployment, and a social adjustment scale score indicative of non-optimal functiong (≥ 3) were considered risk factors, coded as "1", and then tallied. Range of scores 0 (less)-3 (more risk).
Time Frame: 2.5 years
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cross-Sectional: New participants and former participants studied cross-sectionally.
Arm/Group | Cross-Sectional
Number analyzed (Participants) | 151
units on a scale
  Cumulative Adversity Score | 3.24 (2.73)
  Overall Childhood Adversity | 22.41 (29.98)
  Social Adjustment Scale | 2.47 (1.21)
  Psychosocial Risk Factors | 1.03 (0.88)

3. Primary Outcome: Psychosocial Health Risk Factors Correlated With BMI
Description: Correlations of scales with BMI score. Cumulative adversity occurring before age 18 was assessed using a) the Evaluation of Lifetime Stressors, b) SCID, and c) the Adult Attachment Interview. A cumulative adversity sum score was obtained (range 0-13; higher is more adversity). An overall adversity score was created by multiplying the number of childhood adversities × the overall severity of childhood adversity × the overall chronicity of childhood adversity. Scores for overall adversity ranged from 0 to 156 (higher is more adversity). The Social Adjustment Scale is a semi-structured interview assessing functioning in the preceding 2 months and ranges from 1 (excellent adjustment) to 7 (very poor adjustment). Psychosocial risk factors is an index of 1 to 3 (higher is more risk). Health risk score adds smoking, non-optimal drinking (>7/14 drinks/week for women/men), a score in the bottom tertile of the AHEI, and minimal exercise (<6 hours/week)and tallied (scores0-4 with higher worse).
Time Frame: 2.5 years
Measure: Number; unit: Pearson Correlation Coefficients
Arm/Group | Cross-Sectional
Number analyzed (Participants) | 151
Pearson Correlation Coefficients
  Cumulative Adversity Score with BMI | 0.17
  Psychosocial Risk Factors with BMI | 0.23
  Social Adjustment with BMI | -0.17
  Cumulative Adversity Score with Health Risk Factor | 0.14
  Psychosocial Risk Factors with Health Risk Factors | 0.49
  Social Adjustment with Health Risk Factors | 0.45

4. Primary Outcome: Social Adjustment Scale
Description: The Social Adjustment Scale is a semi-structured interview assessing functioning in the preceding 2 months in domains of work (including employment functioning, homemaking and other household functions, and/or student/educational functioning), friendships/leisure, and relationships with extended family. If applicable, relationships with immediate family members (spouse/partner and/or children) are also assessed. The SAS is closely linked to mental health and can be used as a tool for assessing treatment response to psychotropic medications or therapies. Positive adjustment is the ability to carry out each activity/role effectively, deriving satisfaction/support from that domain, whereas poor adjustment reflects maladaptation, dissatisfaction, disengagement, and/or discord. Scores range from 1 (excellent adjustment) to 7 (very poor adjustment). Coding was completed during an audio-recorded interview; 12% were coded for agreement (91%).
Time Frame: 2.5 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cross-Sectional
Number analyzed (Participants) | 151
units on a scale | 2.47 (1.21)

5. Secondary Outcome: Body Mass Index (BMI)
Description: BMI is calculated as weight in kilograms divided by height in meters squared.
Time Frame: cross-sectional
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Cross-Sectional
Number analyzed (Participants) | 151
kg/m^2 | 30.41 (7.22)

6. Secondary Outcome: Health Risk Factors
Description: An index score of health behavior risk factors was created. Any amount of smoking, non-optimal drinking (≥ 7 drinks per week for women; ≥ 14 drinks per week for men), a score in the bottom tertile of the AHEI, and minimal exercise (< 6 metabolic hours per week) were considered risk factors, coded as "1", and then tallied. The range of scores for health risk factors in the current sample was between 0 and 4 health risk factors (where 4 is more risk factors).
Time Frame: cross-sectional
Measure: Mean (Standard Deviation); unit: sum of health risk factors
Arm/Group | Cross-Sectional
Number analyzed (Participants) | 151
sum of health risk factors | 1.33 (1.06)

ADVERSE EVENTS:
Time Frame: at cross-sectional or longitudinal visit
Description: Adverse Events would be those noticed at a visit. As no interventions were given/this is an observational study, no adverse events were expected.
Arm/Group | Cross-Sectional
All-Cause Mortality (participants affected / at risk) | 0/151
Serious Adverse Events (participants affected / at risk) | 0/151
Other Adverse Events (participants affected / at risk) | 0/151

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No